CLINICAL TRIAL: NCT02998645
Title: SOAR, Interventional Phase II Single-arm Study to Assess Efficacy and Safety of Eltrombopag Combined With Cyclosporine as First Line Therapy in Adult Patients With Severe Acquired Aplastic Anemia
Brief Title: Eltrombopag Combined With Cyclosporine as First Line Therapy in Patients With Severe Acquired Aplastic Anemia
Acronym: SOAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETB115E2403; 2016-002814-29 (EudraCT Number)
Record Dates: First submitted 2016-11-04; First posted 2016-12-20 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-02

CONDITIONS: Severe Aplastic Anemia
Keywords: severe acquired aplastic anemia; SAA; first line; eltrombopag; cyclosporine; h-ATG; severe aplastic anemia; aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag + cyclosporine (Experimental): Participants received eltrombopag (orally, 150 mg once daily for non-Asian participants / 100 mg once daily for participants of Asian ancestry) in combination with cyclosporine (orally, 10.0 mg/kg/day in divided doses every 12 hours) for up to 6 months. Thereafter, responders at Month 6 were treated with cyclosporine until Month 24
  Interventions: Drug: eltrombopag; Drug: Cyclosporine

INTERVENTIONS:
Drug: eltrombopag — Film-coated tablets (12.5 mg, 25 mg, 50 mg and 75 mg) administered orally, once daily for up to 6 months. East and Southeast Asian participants were treated with 100 mg once daily, to adjust for the lower apparent clearance of eltrombopag. All other participants were treated with 150 mg once daily.
  Other Names: ETB115
Drug: Cyclosporine — Supplied as oral soft gel capsules. The starting dose was based on body weight at 10.0 mg/kg/day (acceptable rounding range was from 9.5 to 10.5 mg/kg/day) in divided doses every 12 hours. After Day 1, dosing was titrated individually according to therapeutic trough level between 200 and 400 μg/L for 6 months. After 6 months (only for responders at Month 6), tapering of cyclosporine was done as follows:
  * 6-9 months: at the 6 months visit, the dose was reduced by 25% for 3 months
  * 9-12 months: at the 9 months visit, the dose was further reduced by 25% for another 3 months
  * 12-24 months: dose was maintained

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of eltrombopag in combination with cyclosporine alone as first-line therapy on overall hematologic response

DETAILED DESCRIPTION:
This was an interventional phase II, single-arm, multicenter, open-label, study to investigate the efficacy and safety of the combination of eltrombopag and cyclosporine in treatment-naive, adult subjects with severe aplastic anemia (SAA) as first line therapy.

Eligible subjects received eltrombopag and cyclosporine for up to 6 months. Participants who achieved hematologic response any time on or before 6 months were considered as responders; else they were considered as non-responders.

Responders at Month 6 discontinued eltrombopag and started to taper cyclosporine until relapse or Month 24, whichever was early. Responders who relapsed prior to 6 months and non-responders discontinued the treatment at 6 months and were followed-up for 30 days.

Responders who started to taper cyclosporine and relapsed prior to 24 months discontinued cyclosporine and were followed-up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had signed the Informed Consent (ICF) prior to any screening procedures
2. Patient was male/female ≥18 years old at the time of informed consent and able to swallow a tablet.
3. Patient had SAA characterized by:

   1. Bone marrow cellularity <30% (excluding lymphocytes) and
   2. At least two of the following (peripheral blood):

      * Absolute neutrophil count <500/µL
      * Platelet count <20,000/µL
      * Absolute reticulocyte count <60,000/µL
4. Normal ECG defined as the following as determined via the mean of a triplicate ECG

   * Resting heart rate: 50-90 bpm
   * QTcF at screening <450 msec (for male patients), ≤460 msec (for female patients)

Exclusion Criteria:

1. Diagnosis of Fanconi anemia.
2. Evidence of a clonal hematologic bone marrow disorder on cytogenetics by central review
3. Prior immunosuppressive therapy with cyclosporine, alemtuzumab, rabbit or horse ATG and thrombopoietin receptor (TPO-R) agonists.
4. Hypersensitivity to eltrombopag or cyclosporine or their components.
5. AST or ALT >3 x ULN.
6. Serum creatinine, total bilirubin, or alkaline phosphatase >1.5 x ULN.
7. Patient with liver cirrhosis.
8. Patients who were human immune deficiency virus (HIV), hepatitis C virus or hepatitis B surface antigen (HBsAg) positive. HCV-RNA negative patients were allowed to be enrolled.
9. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to consent, be compliant with study procedures, tolerate protocol therapy, or that death within 30 days is likely.
10. Patients with cancer who were not considered cure, were on active chemotherapeutic treatment or who took drugs with hematological effects.
11. Administration of an investigational drug within 30 days or 5 half-lives, whichever was longer, preceding the first dose of study treatment.
12. Pregnancy statements and contraception requirements:

    Pregnancy or nursing (lactating) women Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant (or female partners of male patients), unless they were using highly effective methods of contraception during dosing and for 3 months after stopping medication.
13. Not able to understand the investigation nature of the study or to give informed consent.
14. Clinically significant ECG abnormality including cardiac arrhythmias (e. g. ventricular tachycardia) complete left bundle branch block, high grade atrioventricular block, or inability to determine the QTcF interval on the ECG.
15. Presence of cardiac disease, or family history of idiopathic sudden death or congenital long QT syndrome.
16. Risk factors for Torsades de Pointe including uncorrected hypokalemia or hypomagnesemia, or use of concomitant medication(s) with a known risk to prolong the QT interval that could not be discontinued or replaced by safe alternative medication per www.qtdrugs.org.
17. ECOG performance status of ≥2.
18. Patients under the age of 40 must be referred for consideration of allogeneic bone marrow transplantation (HSCT) if (human leukocyte antigen) HLA matching had been done and a suitable matched sibling donor was available and the patient was willing to undergo transplantation (i.e. patients who did not have a HLA match or were not medically fit, not willing or unable to undergo transplantation were considered for enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Brazil (2):
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Hong Kong, Hong Kong
- India (2):
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Vellore
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BR
  - Novartis Investigative Site, Milan, MI
- Mexico (3):
  - Novartis Investigative Site, Mexico D F, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Puebla City
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Madrid
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scheinberg P, Finelli C, Montano-Figueroa EH, Vallejo C, Norasetthada L, Calado RT, Turgut M, Peffault de Latour R, Kriemler-Krahn U, Haenig J, Clark J, Jang J. Activity and safety of eltrombopag in combination with cyclosporin A as first-line treatment of adults with severe aplastic anaemia (SOAR): a phase 2, single-arm study. Lancet Haematol. 2024 Mar;11(3):e206-e215. doi: 10.1016/S2352-3026(23)00395-2. Epub 2024 Feb 6. PMID 38335978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 20 centers in 9 countries.
Pre-assignment Details: Participants received a combination of eltrombopag and cyclosporine for 6 months (Treatment period 1). Participants who were responders at 6 months were followed-up for cyclosporine tapering until relapse or Month 24 whichever was earlier (Treatment period 2)
Groups:
- Eltrombopag + Cyclosporine: Participants received eltrombopag (orally, 100 mg once daily for East/Southeast Asian participants / 150 mg once daily for all other participants) in combination with cyclosporine (orally, 10.0 mg/kg/day in divided doses every 12 hours) for up to 6 months. Thereafter, responders at Month 6 were treated with cyclosporine until Month 24
Period: Treatment Period 1
Arm/Group | Eltrombopag + Cyclosporine
Started | 54
East/Southeast Asian Ethnicity | 18
Non-East/Southeast Asian Ethnicity | 36
Completed | 35
Not Completed | 19
Not completed — Adverse Event | 6
Not completed — Death | 5
Not completed — Technical Problems | 4
Not completed — Lack of Efficacy | 2
Not completed — Progressive disease | 1
Not completed — Subject/guardian decision | 1
Period: Treatment Period 2
Arm/Group | Eltrombopag + Cyclosporine
Started (Participants who were responders at Month 6) | 21
Completed | 11
Not Completed | 10
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 2
Not completed — Progressive disease | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (17.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Southeast Asian | 11
  East Asian | 7
  West Asian | 5
  Other | 4
  South Asian | 3
  Mixed ethnicity | 1
  Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Hematologic Response Rate by 6 Months
Description: Overall hematologic response rate by 6 months was defined as the percentage of participants with complete response (CR) or partial response (PR) any time on or before 6 months.
  PR was defined as any two of the following parameters at two consecutive measurements at least 7 days apart and no platelet transfusion within 7 days of platelet measurement:
  * Absolute neutrophil count (ANC) >500/μL
  * Platelet count >20 000/μL
  * Reticulocyte count >60 000/μL
  CR was defined as all three parameters meet the following criteria at two consecutive measurements at least 7 days apart and no platelet transfusions within 7 days of platelet measurement and no red blood cell transfusion with 14 days of the hemoglobin measurements:
  * ANC > 1 000/μL
  * Platelet count >100 000/μL
  * Hemoglobin >10 g/L
Time Frame: Up to 6 months
Population: Full Analysis Set (FAS) including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Percentage of participants | 46.3 [32.6 to 60.4]

2. Secondary Outcome: Overall Hematologic Response Rate by 3 Months
Description: Overall hematologic response rate by 3 months was defined as the percentage of participants with CR or PR any time on or before 3 months.
  PR was defined as any two of the following parameters at two consecutive measurements at least 7 days apart and no platelet transfusion within 7 days of platelet measurement:
  * ANC >500/μL
  * Platelet count >20 000/μL
  * Reticulocyte count >60 000/μL
  CR was defined as all three parameters meet the following criteria at two consecutive measurements at least 7 days apart and no platelet transfusions within 7 days of platelet measurement and no red blood cell transfusion with 14 days of the hemoglobin measurements:
  * ANC > 1 000/μL
  * Platelet count >100 000/μL
  * Hemoglobin >10 g/L
Time Frame: Up to 3 months
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Percentage of participants | 40.7 [27.6 to 55.0]

3. Secondary Outcome: Overall Hematologic Response Rate at 12 and 24 Months
Description: Overall hematologic response rate at 12 and 24 months was defined as the percentage of participants with CR or PR at 12 and 24 months respectively.
  PR was defined as any two of the following parameters at two consecutive measurements at least 7 days apart and no platelet transfusion within 7 days of platelet measurement:
  * ANC>500/μL
  * Platelet count >20 000/μL
  * Reticulocyte count >60 000/μL
  CR was defined as all three parameters meet the following criteria at two consecutive measurements at least 7 days apart and no platelet transfusions within 7 days of platelet measurement and no red blood cell transfusion with 14 days of the hemoglobin measurements:
  * ANC > 1 000/μL
  * Platelet count >100 000/μL
  * Hemoglobin >10 g/L
Time Frame: 12 and 24 months
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Percentage of participants
  At 12 months | 18.5 [9.3 to 31.4]
  At 24 months | 18.5 [9.3 to 31.4]

4. Secondary Outcome: Duration of First Hematologic Response
Description: Duration of first hematologic response is the time from the date of the start of first response to the date of first relapse. Relapse is defined as no longer meeting definition of PR or CR. Kaplan-Meier method was used for the analysis. If no relapse occurred, the participant was censored at the date of last contact. Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24. PR was defined as any 2 of the following parameters at 2 consecutive measurements at least 7 days apart and no platelet transfusion within 7 days of platelet measurement:
  * ANC >500/μL
  * Platelet count >20 000/μL
  * Reticulocyte count >60 000/μL.
  CR was defined as all 3 parameters meet the following criteria at 2 consecutive measurements at least 7 days apart and no platelet transfusions within 7 days of platelet measurement and no red blood cell transfusion with 14 days of the hemoglobin measurements:
  * ANC >1 000/μL
  * Platelet count >100 000/μL
  * Hemoglobin >10 g/L
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: All participants in the FAS who achieved hematologic response (either CR or PR) any time on or before the 6 months visit
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 25
Days | 351.0 [99.0 to NA] — NA: Not estimable due to the low number of participants with events

5. Secondary Outcome: Relapse Rate by 6 and 24 Months
Description: Relapse was defined as no longer meeting the definition of PR (and not CR). Relapse rate by 6 months and 24 was defined as the percentage of responders by 6 months who relapsed prior to 6 months or prior to 24 months respectively. Responders by 6 months were participants who achieved CR or PR any time on or before 6 months. Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
  PR: any 2 of the following parameters at 2 consecutive measurements at least 7 days apart and no platelet transfusion within 7 days of platelet measurement:
  * ANC>500/μL
  * Platelet count>20 000/μL
  * Reticulocyte count>60 000/μL.
  CR: all 3 parameters meet the following criteria at 2 consecutive measurements at least 7 days apart and no platelet transfusions within 7 days of platelet measurement and no red blood cell transfusion with 14 days of the hemoglobin measurements:
  * ANC>1 000/μL
  * Platelet count>100 000/μL
  * Hemoglobin>10 g/L
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 25
Percentage of participants
  By 6 months | 32.0 [14.9 to 53.5]
  By 24 months | 44.0 [24.4 to 65.1]

6. Secondary Outcome: Percentage of Participants With Evolution to Myelodysplasia, Paroxysmal Nocturnal Hemoglobinuria (PNH) and Leukemia
Description: The percentage of participants with evolution to myelodysplasia, PNH and acute leukemia occurring at any time during the study. Clonal evolution to myelodysplasia was defined as a new marrow cytogenic abnormality with or without characteristic dysplastic marrow findings. Clonal evolution to leukemia was defined as greater than 20% peripheral blood and/or marrow blasts. Clonal evolution to paroxysmal nocturnal hemoglobinuria (PNH) was defined as a clone at baseline < 10% that rose to greater than 50% on study.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Percentage of participants | 0

7. Secondary Outcome: Percentage of Participants Who Were Red Blood Cells (RBC) Transfusion Independent
Description: Percentage of participants who were RBC transfusion independent at least once by 6 months and by 24 months (responders only). Independence was defined as no RBC transfusion for at least 56 days.
  Results are presented for responders and non-responders. If any participant achieved hematologic response (either CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Participants
  Day 1 to 6 months- Responders: number analyzed (Participants) | 25
  Day 1 to 6 months- Responders | 17
  Day 1 to 24 months- Responders: number analyzed (Participants) | 25
  Day 1 to 24 months- Responders | 20
  Day 1 to 6 months- Non-Responders: number analyzed (Participants) | 29
  Day 1 to 6 months- Non-Responders | 5

8. Secondary Outcome: Percentage of Participants Who Were Platelet Transfusion Independent
Description: Percentage of participants who were platelet transfusion independent at least once by 6 months and by 24 months (responders only). Independence was defined as no platelet transfusion for at least 28 days.
  Results are presented for responders and non-responders. If any participant achieved hematologic response (either CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine).
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Participants
  Day 1 to 6 months- Responders: number analyzed (Participants) | 25
  Day 1 to 6 months- Responders | 25
  Day 1 to 24 months- Responders: number analyzed (Participants) | 25
  Day 1 to 24 months- Responders | 25
  Day 1 to 6 months- Non-responders: number analyzed (Participants) | 29
  Day 1 to 6 months- Non-responders | 13

9. Secondary Outcome: Longest Duration of Transfusion Independence (Platelet or RBC)
Description: Longest duration of transfusion independence (platelet or RBC) by 6 months and by 24 months (responders only). Transfusion independence was defined as no transfusions required in at least a 28-day period for platelet transfusion and at least 56-day period for RBC transfusion. The duration of the longest interval with transfusion independence was summarized using Kaplan-Meier analysis.
  Results are presented for responders and non-responders. If any participant achieved hematologic response (either CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24
Time Frame: Up to 6 months (non-responders at Month 6) and up to 24 months (responders at Month 6)
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Days
  Day 1 to 6 months- Responders: number analyzed (Participants) | 25
  Day 1 to 6 months- Responders | NA [NA to NA] — NA: not estimable due to the low number of participants with events
  Day 1 to 24 months- Responders: number analyzed (Participants) | 25
  Day 1 to 24 months- Responders | NA [498.0 to NA] — NA: not estimable due to the low number of participants with events
  Day 1 to 6 months- Non-Responders: number analyzed (Participants) | 29
  Day 1 to 6 months- Non-Responders | 87.0 [48.0 to NA] — NA: not estimable due to the low number of participants with events

10. Secondary Outcome: Change From Baseline in Scores of Functional Assessment of Cancer Therapy - General (FACT-G) Patient Reported Outcome
Description: The FACT-G consists of 27-items divided into 4 domains (physical well-being, social well-being, emotional and functional well-being). All items of the FACT-G use a 5 point scale ranging from 0 to 4 with a 0 rating being "not at all" and a 4 rating being "very much". Total FACT-G score is the sum of physical well-being score, social well-being score, emotional well-being score and functional well-being score. Score ranges from 0 to 108, with higher scores indicating better quality of life (QoL). A positive change from baseline indicates improvement in the QoL.
  Results are presented for responders and non-responders. If any participant achieved hematologic response (either CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
Time Frame: Baseline, every 2 weeks from Week 2 to Week 24 or End of Treatment Period 1 (for all participants); and at Week 38, Week 53, Month 24 or End of Treatment Period 2 (for responders at Month 6 only)
Population: FAS including all subjects who received at least one dose of study treatment (eltrombopag or cyclosporine). Only participants with an evaluable baseline visit and at least one evaluable post-baseline visit were included in the analysis. Number analyzed are the number of participants with data available for analysis at the given category.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Score on a scale
  Week 2 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 2 (Treatment period 1) - Responders | -2.0 [-26 to 30]
  Week 4 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 4 (Treatment period 1) - Responders | -3.0 [-22 to 23]
  Week 6 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 6 (Treatment period 1) - Responders | -0.3 [-48 to 30]
  Week 8 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 8 (Treatment period 1) - Responders | 0.0 [-25 to 30]
  Week 10 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 10 (Treatment period 1) - Responders | -1.3 [-43 to 33]
  Week 12 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 12 (Treatment period 1) - Responders | 0.8 [-40 to 30]
  Week 14 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 14 (Treatment period 1) - Responders | 1.0 [-44 to 29]
  Week 16 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 16 (Treatment period 1) - Responders | -2.0 [-51 to 35]
  Week 18 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 18 (Treatment period 1) - Responders | 3.0 [-41 to 37]
  Week 20 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 20 (Treatment period 1) - Responders | -1.0 [-46 to 41]
  Week 22 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 22 (Treatment period 1) - Responders | 1.0 [-43 to 39]
  Week 24 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 24 (Treatment period 1) - Responders | 1.8 [-46 to 35]
  Week 26 (Treatment period 1) - Responders: number analyzed (Participants) | 19
  Week 26 (Treatment period 1) - Responders | 1.0 [-51 to 38]
  End of treatment period 1 - Responders: number analyzed (Participants) | 22
  End of treatment period 1 - Responders | -1.0 [-51 to 38]
  Week 38 (Treatment period 2)- Responders: number analyzed (Participants) | 15
  Week 38 (Treatment period 2)- Responders | 5.7 [-43 to 47]
  Week 53 (Treatment period 2)- Responders: number analyzed (Participants) | 15
  Week 53 (Treatment period 2)- Responders | 4.0 [-46 to 42]
  Month 24 (Treatment period 2)- Responders: number analyzed (Participants) | 10
  Month 24 (Treatment period 2)- Responders | 22.0 [-50 to 84]
  End of treatment period 2 - Responders: number analyzed (Participants) | 8
  End of treatment period 2 - Responders | 13.5 [-5 to 47]
  Week 2 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 28
  Week 2 (Treatment period 1) - Non-Responders | -0.3 [-34 to 21]
  Week 4 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 23
  Week 4 (Treatment period 1) - Non-Responders | -1.0 [-42 to 22]
  Week 6 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 6 (Treatment period 1) - Non-Responders | -3.6 [-45 to 17]
  Week 8 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 8 (Treatment period 1) - Non-Responders | 1.5 [-36 to 99]
  Week 10 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 10 (Treatment period 1) - Non-Responders | -0.9 [-27 to 25]
  Week 12 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 12 (Treatment period 1) - Non-Responders | -0.3 [-54 to 26]
  Week 14 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 14 (Treatment period 1) - Non-Responders | -0.3 [-39 to 28]
  Week 16 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 16 (Treatment period 1) - Non-Responders | 0.3 [-50 to 23]
  Week 18 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 18 (Treatment period 1) - Non-Responders | -2.6 [-45 to 19]
  Week 20 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 14
  Week 20 (Treatment period 1) - Non-Responders | -1.5 [-44 to 22]
  Week 22 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 15
  Week 22 (Treatment period 1) - Non-Responders | -1.0 [-45 to 12]
  Week 24 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 14
  Week 24 (Treatment period 1) - Non-Responders | 2.7 [-30 to 18]
  Week 26 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 11
  Week 26 (Treatment period 1) - Non-Responders | -2.7 [-25 to 24]
  End of treatment period 1 - Non-Responders: number analyzed (Participants) | 19
  End of treatment period 1 - Non-Responders | -2.0 [-30 to 24]

11. Secondary Outcome: Change From Baseline in Scores of FACT - Thrombocytopenia 18 (FACT-TH18) Patient Reported Outcome
Description: The FACT-TH18 is comprised of FACT-G and a thrombocytopenia specific questionnaire. FACT-G consists of 27-items divided into 4 domains (physical, social, emotional and functional well-being). FACT-TH18 has 18 additional items which asks the patient to rate degree of thrombocytopenia. All items of the FACT-TH18 use a 5 point scale ranging from 0 to 4, with 0 = "not at all" and 4 = "very much". Total FACT-TH18 score is the sum of physical, social, emotional and functional well-being scores, and thrombocytopenia subscale. Score ranges from 0 to 180, with higher scores indicating better QoL. A positive change from baseline indicates improvement in the QoL. Results are presented for responders and non-responders. If any participant achieved hematologic response (CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders. Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Score on a scale
  Week 2 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 2 (Treatment period 1) - Responders | 2.3 [-43 to 43]
  Week 4 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 4 (Treatment period 1) - Responders | -1.5 [-37 to 54]
  Week 6 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 6 (Treatment period 1) - Responders | 8.4 [-62 to 70]
  Week 8 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 8 (Treatment period 1) - Responders | 9.0 [-34 to 66]
  Week 10 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 10 (Treatment period 1) - Responders | 3.4 [-44 to 73]
  Week 12 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 12 (Treatment period 1) - Responders | 9.3 [-45 to 69]
  Week 14 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 14 (Treatment period 1) - Responders | 6.4 [-45 to 63]
  Week 16 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 16 (Treatment period 1) - Responders | 7.8 [-47 to 68]
  Week 18 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 18 (Treatment period 1) - Responders | 13.9 [-46 to 77]
  Week 20 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 20 (Treatment period 1) - Responders | 11.8 [-48 to 81]
  Week 22 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 22 (Treatment period 1) - Responders | 13.5 [-46 to 81]
  Week 24 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 24 (Treatment period 1) - Responders | 14.5 [-48 to 72]
  Week 26 (Treatment period 1) - Responders: number analyzed (Participants) | 19
  Week 26 (Treatment period 1) - Responders | 18.2 [-57 to 72]
  End of treatment period 1 - Responders: number analyzed (Participants) | 22
  End of treatment period 1 - Responders | 13.9 [-57 to 72]
  Week 38 (Treatment period 2)- Responders: number analyzed (Participants) | 15
  Week 38 (Treatment period 2)- Responders | 21.7 [-50 to 88]
  Week 53 (Treatment period 2)- Responders: number analyzed (Participants) | 13
  Week 53 (Treatment period 2)- Responders | 22.0 [-50 to 84]
  Month 24 (Treatment period 2)- Responders: number analyzed (Participants) | 10
  Month 24 (Treatment period 2)- Responders | 35.7 [5 to 95]
  End of treatment period 2 - Responders: number analyzed (Participants) | 8
  End of treatment period 2 - Responders | 6.9 [-55 to 35]
  Week 2 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 28
  Week 2 (Treatment period 1) - Non-Responders | 0.6 [-78 to 39]
  Week 4 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 23
  Week 4 (Treatment period 1) - Non-Responders | 2.1 [-77 to 45]
  Week 6 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 6 (Treatment period 1) - Non-Responders | -1.5 [-97 to 42]
  Week 8 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 8 (Treatment period 1) - Non-Responders | 2.0 [-54 to 43]
  Week 10 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 10 (Treatment period 1) - Non-Responders | 5.2 [-22 to 41]
  Week 12 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 12 (Treatment period 1) - Non-Responders | 1.8 [-101 to 49]
  Week 14 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 14 (Treatment period 1) - Non-Responders | 2.8 [-64 to 41]
  Week 16 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 16 (Treatment period 1) - Non-Responders | 2.1 [-98 to 38]
  Week 18 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 18 (Treatment period 1) - Non-Responders | 0.5 [-78 to 27]
  Week 20 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 14
  Week 20 (Treatment period 1) - Non-Responders | 2.4 [-68 to 43]
  Week 22 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 15
  Week 22 (Treatment period 1) - Non-Responders | -1.3 [-67 to 39]
  Week 24 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 14
  Week 24 (Treatment period 1) - Non-Responders | 0.7 [-31 to 43]
  Week 26 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 11
  Week 26 (Treatment period 1) - Non-Responders | -1.4 [-24 to 41]
  End of treatment period 1 - Non-Responders: number analyzed (Participants) | 19
  End of treatment period 1 - Non-Responders | -1.4 [-27 to 41]

12. Secondary Outcome: Change From Baseline in Scores of Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT- Fatigue) Patient Reported Outcome
Description: The FACIT- Fatigue is a 13-item fatigue subscale that asks the patient to rate their degree of tiredness, weakness and fatigue. All items of the FACIT-Fatigue use a 5-point scale ranging from 0 to 4 with a 0 rating being "not at all" and a 4 rating being "very much". Total score ranges from 0 to 52. Negatively worded items were reverse scored before summing so that higher total scores indicate less fatigue. A positive change from baseline indicates improvement.
  Results are presented for responders and non-responders. If any participant achieved hematologic response (either CR or PR) any time on or before 6 months, they were considered as responders, else they were considered as non-responders.
  Only participants who achieved hematologic response of CR or PR at Month 6 were followed up until Month 24.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 54
Score on a scale
  Week 2 (Treatment period 1) - Responders: number analyzed (Participants) | 23
  Week 2 (Treatment period 1) - Responders | 3.0 [-13 to 34]
  Week 4 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 4 (Treatment period 1) - Responders | 2.0 [-16 to 22]
  Week 6 (Treatment period 1) - Responders: number analyzed (Participants) | 23
  Week 6 (Treatment period 1) - Responders | 4.0 [-22 to 32]
  Week 8 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 8 (Treatment period 1) - Responders | 6.0 [-7 to 29]
  Week 10 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 10 (Treatment period 1) - Responders | 4.5 [-11 to 30]
  Week 12 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 12 (Treatment period 1) - Responders | 5.5 [-11 to 31]
  Week 14 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 14 (Treatment period 1) - Responders | 6.5 [-5 to 26]
  Week 16 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 16 (Treatment period 1) - Responders | 6.0 [-5 to 28]
  Week 18 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 18 (Treatment period 1) - Responders | 7.0 [-5 to 28]
  Week 20 (Treatment period 1) - Responders: number analyzed (Participants) | 21
  Week 20 (Treatment period 1) - Responders | 6.0 [-5 to 29]
  Week 22 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 22 (Treatment period 1) - Responders | 6.0 [-8 to 33]
  Week 24 (Treatment period 1) - Responders: number analyzed (Participants) | 22
  Week 24 (Treatment period 1) - Responders | 6.0 [-5 to 29]
  Week 26 (Treatment period 1) - Responders: number analyzed (Participants) | 19
  Week 26 (Treatment period 1) - Responders | 7.0 [-9 to 32]
  End of treatment period 1 - Responders: number analyzed (Participants) | 22
  End of treatment period 1 - Responders | 6.0 [-9 to 32]
  Week 38 (Treatment period 2)- Responders: number analyzed (Participants) | 15
  Week 38 (Treatment period 2)- Responders | 6.0 [-8 to 33]
  Week 53 (Treatment period 2)- Responders: number analyzed (Participants) | 13
  Week 53 (Treatment period 2)- Responders | 8.0 [-2 to 41]
  Month 24 (Treatment period 2)- Responders: number analyzed (Participants) | 11
  Month 24 (Treatment period 2)- Responders | 9.0 [1 to 31]
  End of treatment period 2 - Responders: number analyzed (Participants) | 8
  End of treatment period 2 - Responders | 11.5 [-5 to 42]
  Week 2 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 28
  Week 2 (Treatment period 1) - Non-Responders | -0.5 [-23 to 19]
  Week 4 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 23
  Week 4 (Treatment period 1) - Non-Responders | -2.0 [-38 to 20]
  Week 6 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 6 (Treatment period 1) - Non-Responders | 0.0 [-43 to 18]
  Week 8 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 20
  Week 8 (Treatment period 1) - Non-Responders | -1.0 [-27 to 14]
  Week 10 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 10 (Treatment period 1) - Non-Responders | 0.5 [-25 to 16]
  Week 12 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 17
  Week 12 (Treatment period 1) - Non-Responders | -1.0 [-42 to 15]
  Week 14 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 14 (Treatment period 1) - Non-Responders | -1.5 [-43 to 16]
  Week 16 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 16 (Treatment period 1) - Non-Responders | -0.5 [-46 to 15]
  Week 18 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 16
  Week 18 (Treatment period 1) - Non-Responders | -6.0 [-43 to 15]
  Week 20 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 15
  Week 20 (Treatment period 1) - Non-Responders | -6.0 [-45 to 22]
  Week 22 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 15
  Week 22 (Treatment period 1) - Non-Responders | -4.0 [-45 to 15]
  Week 24 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 14
  Week 24 (Treatment period 1) - Non-Responders | -7.0 [-19 to 12]
  Week 26 (Treatment period 1) - Non-Responders: number analyzed (Participants) | 11
  Week 26 (Treatment period 1) - Non-Responders | -8.0 [-19 to 15]
  End of treatment period 1 - Non-Responders: number analyzed (Participants) | 19
  End of treatment period 1 - Non-Responders | -4.0 [-19 to 15]

13. Secondary Outcome: Pharmacokinetic Parameter- Cmax of Eltrombopag When Combined With Cyclosporine
Description: Cmax is the observed maximum plasma concentration following administration. The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 microgram/milliliter (ug/mL). Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose and 2, 4, 6 and 8 hours post-dose.
Population: Participants in the Pharmacokinetic Analysis Set (PAS) including participants who provided at least one evaluable PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 44
microgram/milliliter (ug/mL)
  East/Southeast Asian ethnicity: number analyzed (Participants) | 18
  East/Southeast Asian ethnicity | 29.1 (43.5)
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 26
  Non-East/Southeast Asian ethnicity | 38.7 (38.0)

14. Secondary Outcome: Pharmacokinetic Parameter-AUClast of Eltrombopag When Combined With Cyclosporine
Description: AUClast is the area under the curve calculated to the last quantifiable concentration point (Tlast). The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 ug/mL. Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose and 2, 4, 6 and 8 hours post-dose
Population: Participants in the Pharmacokinetic Analysis Set (PAS) including participants who provided at least one evaluable PK concentration. Only participants with an evaluable PK parameter (Cmax) were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*ug/mL)
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 44
hour*microgram/milliliter (h*ug/mL)
  East/Southeast Asian ethnicity: number analyzed (Participants) | 18
  East/Southeast Asian ethnicity | 583 (38.3)
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 26
  Non-East/Southeast Asian ethnicity | 702 (59.9)

15. Secondary Outcome: Pharmacokinetic Parameter- AUCtau of Eltrombopag When Combined With Cyclosporine
Description: AUCtau is the area under the curve calculated to the end of the dosing interval (tau). The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 ug/mL. Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose and 2, 4, 6 and 8 hours post-dose
Population: Participants in the Pharmacokinetic Analysis Set (PAS) including participants who provided at least one evaluable PK concentration. Only participants with an evaluable PK parameter (AUCtau) were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*ug/mL)
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 18
hour*microgram/milliliter (h*ug/mL)
  East/Southeast Asian ethnicity: number analyzed (Participants) | 8
  East/Southeast Asian ethnicity | 686 (32.4)
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 10
  Non-East/Southeast Asian ethnicity | 727 (33.0)

16. Secondary Outcome: Pharmacokinetic Parameter- Ctrough of Eltrombopag When Combined With Cyclosporine
Description: Ctrough is the pre-dose plasma concentration. The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 ug/mL. Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose
Population: Participants in the Pharmacokinetic Analysis Set (PAS) including participants who provided at least one evaluable PK concentration. Only participants with an evaluable PK parameter (Ctrough) were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 45
microgram/milliliter (ug/mL)
  East/Southeast Asian ethnicity: number analyzed (Participants) | 18
  East/Southeast Asian ethnicity | 19.3 (45.3)
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 27
  Non-East/Southeast Asian ethnicity | 27.2 (44.1)

17. Secondary Outcome: Pharmacokinetic Parameter- Tmax of Eltrombopag When Combined With Cyclosporine
Description: Tmax is the time to reach peak or maximum concentration. The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 ug/mL. Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose and 2, 4, 6 and 8 hours post-dose
Population: Participants in the Pharmacokinetic Analysis Set (PAS) including participants who provided at least one evaluable PK concentration. Only participants with an evaluable PK parameter (Tmax) were included in the analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 44
Hours
  East/Southeast Asian ethnicity: number analyzed (Participants) | 18
  East/Southeast Asian ethnicity | 5.79 [1.93 to 8.00]
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 26
  Non-East/Southeast Asian ethnicity | 3.75 [0.00 to 8.00]

18. Secondary Outcome: Pharmacokinetic Parameter- CLss/F of Eltrombopag When Combined With Cyclosporine
Description: CLss/F is the apparent systemic (or total body) clearance at steady state from plasma. The plasma samples from all participants were assayed for eltrombopag concentrations using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS). The lower limit of quantitation (LLOQ) was 0.1 ug/mL. Concentration values below the LLOQ were reported as zero, and missing samples were labeled accordingly. Results are reported by ethnicity: East/Southeast Asian participants received eltrombopag planned dose of 100mg/day and all other participants received eltrombopag planned dose of 150mg/day.
Time Frame: Week 2 at pre-dose and 2, 4, 6 and 8 hours post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour (mL/h)
Arm/Group | Eltrombopag + Cyclosporine
Number analyzed (Participants) | 18
milliliter/hour (mL/h)
  East/Southeast Asian ethnicity: number analyzed (Participants) | 8
  East/Southeast Asian ethnicity | 146 (32.4)
  Non-East/Southeast Asian ethnicity: number analyzed (Participants) | 10
  Non-East/Southeast Asian ethnicity | 206 (33.0)

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to 30 days after last dose of study medication, assessed up to 25 months
Arm/Group | Eltrombopag + Cyclosporine
All-Cause Mortality (participants affected / at risk) | 8/54
Serious Adverse Events (participants affected / at risk) | 27/54
Other Adverse Events (participants affected / at risk) | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag + Cyclosporine (N=54)
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Cardiac arrest (Cardiac disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Gastric dysplasia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 2
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Prostatic abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag + Cyclosporine (N=54)
Palpitations (Cardiac disorders) | 3
Retinal haemorrhage (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 7
Gingival hypertrophy (Gastrointestinal disorders) | 6
Mouth haemorrhage (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Odynophagia (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 4
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 4
Oral candidiasis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 10
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 22
Blood creatinine increased (Investigations) | 10
Neutrophil count decreased (Investigations) | 3
SARS-CoV-2 test positive (Investigations) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Iron overload (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT02998645/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02998645/SAP_001.pdf